CLINICAL TRIAL: NCT00588536
Title: Study of Sequential Administration of Oral 6-Thioguanine After Methotrexate in Patients With Langerhans Cell in Histiocytosis (LCH)
Brief Title: Study of Sequential Administration of Oral 6-Thioguanine After Methotrexate in Patients With LCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 94-132
Record Dates: First submitted 2007-12-26; First posted 2008-01-08 (Estimated); Results first posted 2015-05-04 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Langerhans Cell Histiocytosis
Keywords: Langerhans Cell Histiocytosis; LCH; 6-Thioguanine; 6-TG; Methotrexate; MTX; 94-132
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell | interventions — Methotrexate; Thioguanine; Leucovorin

ARMS (1):
- 1 (Experimental): MTX, 6-TG, Leucovorin
  Interventions: Drug: Methotrexate; Drug: 6-Thioguanine; Drug: Leucovorin Calcium

INTERVENTIONS:
Drug: Methotrexate — MTX 30mg/m2 (or 1mg/kg for infants) orally, given in three equally divided doses at 0,8, and 16hrs
  Other Names: MTX
Drug: 6-Thioguanine — 6-TG 300mg/m2 (or 10mg/kg for infants) orally, given in one dose.
  Other Names: 6-TG
Drug: Leucovorin Calcium — 5mg orally at 36,48, and 60hrs (or 12 hrs after the dose of 6-TG and then every 12 hrs for a total of 3 doses)

SUMMARY:
The objective of this study is to determine the incidence of complete and partial response and the duration of response in patients with Langerhans Cell Histiocytosis (LCH) treated with sequential administration of oral 6-Thioguanine (6-TG) after Methotrexate (MTX).

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologic proof of LCH who have multifocal or multisystem disease involvement.
* Patients must have a life expectancy of at least 8 weeks.
* All patients must have ECOG performance level rating of-< 2.
* Patients or their parents (guardian) must sign an informed consent indicating that they are aware of the investigational nature of the study, using commercially available drugs.
* Patients must have recovered from the toxic effects of prior therapy before entering this study or at least 2 weeks should have elapsed since the end of last course of chemotherapy.
* Patients must have adequate liver function (bilirubin _< 2.0 mg/dl, SGOT less than 1.5 times normal (unless it is due to disease), adequate renal function (creatinine <_ 1.5 mg/dl, creatinine clearance >_ 60 ml/min/1.73 m2) and normal electrolytes.
* Patients should have a granulocyte count > 500/uL and a platelet count >_ 100,000/uL (unless due to disease involvement of the bone marrow).
* Male and female patients of child-bearing age should use effective methods of contraception, if sexually active.

Exclusion Criteria:

* Patients with active infections or significant medical conditions other than their disease (LCH) shall be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 1995-01; Primary Completion 2008-07 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Trippett, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual: 01/10/1995 Protocol Closed to Accrual: 07/25/2006 Primary Completion Date (if applicable): 06/09/2009 Recruitment Location is the medical clinic
Groups:
- MTX, 6-TG and Leucovorin: Methotrexate: MTX 30mg/m2 (or 1mg/kg for infants) orally, given in three equally divided doses at 0,8, and 16hrs
  6-Thioguanine: 6-TG 300mg/m2 (or 10mg/kg for infants) orally, given in one dose.
  Leucovorin Calcium: 5mg orally at 36,48, and 60hrs (or 12 hrs after the dose of 6-TG and then every 12 hrs for a total of 3 doses)
Period: Overall Study
Arm/Group | MTX, 6-TG and Leucovorin
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MTX, 6-TG and Leucovorin
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Determine the Incidence of Complete and Partial Response and the Duration of Response in Patients With Langerhans Cell Histiocytosis (LCH) Treated With Sequential Administration of Oral 6-TG After MTX.
Time Frame: Conclusion of the study
Measure: Number; unit: participants
Arm/Group | MTX, 6-TG and Leucovorin
Number analyzed (Participants) | 5
participants
  Complete Response | 2
  Stable Disease | 1
  Progression of Disease | 2

ADVERSE EVENTS:
Arm/Group | MTX, 6-TG and Leucovorin
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MTX, 6-TG and Leucovorin (N=5)
Fever (General disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MTX, 6-TG and Leucovorin (N=5)
Abdominal pain/cramping (Gastrointestinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Creatinine increased (Investigations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (10)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
White blood cell decreased (Investigations) | 2 (4)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 2 (9)
Rash desquamation (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes